CLINICAL TRIAL: NCT01066221
Title: Comparative Study of Enzyme Immunoassays:Techlab Toxins A&B, C Diff Quick Check for Glutamate Dehydrogenase (GDH);3 PCRs,and Cytotoxin Assay (CTA) for the Detection of Clostridium Difficile Toxin in Adult Stool Specimens
Brief Title: Comparative Study of Three Different Testing Mechanisms for Clostridium Difficile
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Christine Lee, MD, McMaster University
Organization: McMaster University (Other)
Other Study IDs: 2010-001
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2010-02

CONDITIONS: Clostridium Difficile
Keywords: clostridium difficile

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clostridium difficile patients: observational study

SUMMARY:
The purpose of this study is to establish which of the following tests perform best in diagnosing clostridium difficile. PCR, Enzyme Immunoassays (EIA) and C. difficile cytotoxin assay (CTA).

DETAILED DESCRIPTION:
This comparative study will be carried out in the hospital microbiology laboratory of a tertiary academic health center, St. Joseph's Healthcare (SJH) affiliated with McMaster University, Hamilton, ON on 500 individual stool samples from patients greater than 12 months of age to determine an efficacy of distinction between current gold standard and other methods of testing for Clostridium difficile. This study is required to find a faster test for diagnosis of CDI in order to facilitate prompt treatment and reduce the complications of CDI. Identification of infected cases will lead to the enforcement of infection control measures and thereby prevent spread to other susceptible children. This is turn will reduce costs, length of stay, morbidity, and mortality from CDI if instituted correctly.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 12 months of age
* Having diarrhea

Exclusion Criteria:

* Inadequate volume of sample to perform all three diagnostic tests (less than 3mL
* Formed stools

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hamilton Regional Laboratory Medicine Program - patients with clostridium difficile
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To establish the performances of the three testing assays to see which one is the best. | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada